CLINICAL TRIAL: NCT04723459
Title: Nano-Ivermectin Impregnated Masks Versus Ordinary Surgical Masks in Prevention of Covid-19 Among Healthy Contacts and Medical Staff
Brief Title: Efficacy of Nano-Ivermectin Impregnated Masks in Prevention of Covid-19 Among Healthy Contacts and Medical Staff
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Zaky Aref, ass.professor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SVU MED CIT0 23 4 21 1 121
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Covid-19
Keywords: Covid-19; antiviral mask; nano ivermectin
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin mask group (Active Comparator): Contacts who will use ivermectin masks
  Interventions: Other: ivermectin impregnated mask
- ordinary mask group (No Intervention): Contacts who will use regular masks

INTERVENTIONS:
Other: ivermectin impregnated mask — mask with ivermectin nano solution
  Arms: Ivermectin mask group

SUMMARY:
Antiviral efficacy of Ivermectin against Covid-19 in vitro was stated by many stusies all over the world with decreased effecacy in vivo so ,usage of masks impregnated into nano Ivermectin solution will theoretically increase the protective action of the ordinary masks

DETAILED DESCRIPTION:
Antiviral effecacy of Ivermectin against Covid-19 in vitro was stated by many stusies all over the world with decreased effecacy in vivo so ,usage of masks impregnated into nano Ivermectin solution will theoretically increase the protective action of the ordinary masks this study is a trial for evaluation of adding a proved antiviral material to the mask and to compare between the protective value of this mask and the ordinary one.

ELIGIBILITY:
Inclusion Criteria:

* health care personells and family contact of confirmed COVID-19 cases.

Exclusion Criteria:

* refusal of participate to use the masks.
* pregnancy or lactation known hypersensitivity to ivermectin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-23 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-03-28 (Estimated)

PRIMARY OUTCOMES:
Number of persons in each group who Complain of any suspected Symptoms | within 14 days after enrollement
  ( Fever, Myalgia ,Cough, Sore Throat, Diarrhea, Shortness of Breath)

SECONDARY OUTCOMES:
Number of persons in each group who are diagnosed as COVID-19 patients | within 21 days after enrollement
  swab test

CONTACTS AND LOCATIONS:
Locations (1):
- Zaky Aref, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- See also: Related Info — https://druginfo.nlm.nih.gov/drugportal/name/Ivermectin